CLINICAL TRIAL: NCT00552994
Title: A Danish Prospective Randomized Multicenter Comparison of the Xience V and the Cypher Select+ Stents in Unselective Patients With Diabetes Mellitus. An Intravascular Ultrasound Study.
Brief Title: Comparison of Coronary Xience V and the Cypher Select+ Stents in Diabetic Patients
Acronym: DIABEDES IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Lisette Okkels Jensen, Odense University Hospital, Denmark
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IVUS-20070043
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitus
Keywords: Drug eluting stent; Diabetics; Intravascular ultrasound; Pathophysiologic (neointimal hyperplasia and peri-stent remodeling)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cypher Select plus stent
  Interventions: Device: Cypher Select plus
- 2 (Active Comparator): Xience V stent
  Interventions: Device: Xience V stent

INTERVENTIONS:
Device: Cypher Select plus — Drug eluting stent
  Arms: 1
Device: Xience V stent — Drug eluting stent
  Arms: 2

SUMMARY:
In stent neointimal hyperplasia may be less in the Cypher select plus stent compared to the Xience V stent in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients treated with one or more drug eluting stents in the coronary arteries at one of the 5 heart centres in Denmark (Gentofte, Rigshospitalet, Odense, Skejby, Aalborg) can be included in the study.

Exclusion Criteria:

* The patient will not participate
* The patient participates in other randomised stent studies
* Expected survival < 1 year
* Allergy to Aspirin, Clopidogrel or Ticlopidine
* Allergy to Sirolimus or ABT-578

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
In stent neointimal hyperplasia | Within 10 months

SECONDARY OUTCOMES:
Peri-stent remodeling - Edge response to Cypher Select plus and Xience V stent - Malapposition - Angiographic late lumen loss | Within 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Thayssen, MD DMSci, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Antonsen L, Maeng M, Thayssen P, Christiansen EH, Hansen KN, Kaltoft A, Hansen HS, Thuesen L, Lassen JF, Jensen LO. Intimal hyperplasia and vascular remodeling after everolimus-eluting and sirolimus-eluting stent implantation in diabetic patients: the randomized Diabetes and Drug-Eluting Stent (DiabeDES) IV Intravascular Ultrasound trial. Catheter Cardiovasc Interv. 2014 May 1;83(6):864-72. doi: 10.1002/ccd.25180. Epub 2013 Sep 30. PMID 23996918